CLINICAL TRIAL: NCT06365619
Title: Phase II Study of Neoadjuvant Ipilimumab/Nivolumab for Patients With Recurrent, High Risk, Resectable Melanoma
Brief Title: Neoadjuvant Ipilimumab/Nivolumab for Patients With Recurrent, High Risk, Resectable Melanoma
Acronym: NeoRelapse
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI168525
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment: All Patients (Experimental): Neoadjuvant Ipilimumab and Nivolumab
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — Two cycles of neoadjuvant ipilimumab prior to surgical resection.
Drug: Nivolumab — two cycles of neoadjuvant nivolumab prior to surgical resection.

SUMMARY:
The goal of this clinical trial is to study the impact of Neoadjuvant ipilimumab and nivolumab for melanoma patients that had recurrence during or after adjuvant anti-PD-1 therapy.

Participants will receive 2 cycles of treatment prior to their standard of care surgery. After surgery participants will receive standard of care adjuvant therapy and be followed for response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years.
* Histologically confirmed Stage IIIB-D or Stage IV recurrent metastatic melanoma that is resectable or borderline resectable as determined by a Surgical Oncologist.
* Recurrent disease at eligibility must have been confirmed with biopsy while receiving or within 3 months of completion of adjuvant anti-PD1 therapy.
* ECOG Performance Status ≤ 1.
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥ 1500/mm3
    * Platelet count ≥ 100,000/mm3
    * Hemoglobin ≥ 10 g/dL
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN ----Subjects with liver metastases will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.
  * Renal:

    * Estimated creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula:
* For subjects of childbearing potential: Negative pregnancy test or evidence of post-menopausal status or evidence of permanent surgical sterilization. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Subjects < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
  * Subjects ≥ 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago
* Subjects of childbearing potential and subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.3.1.
* Subject has adequate archival tissue or agrees to undergo a fresh tissue biopsy if sufficient archival tissue is unavailable.
* Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy per the treating investigator.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Receiving other investigational agents currently or within 28 days of study treatment.
* Prior systemic anti-cancer therapy ≤ 14 days or within five half-lives prior to starting study treatment, whichever is shorter.
* Prior radiotherapy 45 days prior to the first dose of study treatment.
* Major surgery 4 weeks prior to starting study drug or who have not fully recovered from major surgery.
* Active infection requiring the use of systemic antibiotics.
* Systemic steroid therapy greater than physiologic equivalent (10mg prednisone/day) or any other form of systemic immunosuppressive therapy within 7 days prior to registration.
* Active secondary malignancy, unless the malignancy is not expected to interfere with the evaluation of safety
* Known brain metastases or cranial epidural disease.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  --Cardiovascular disorders:
  * Congestive heart failure New York Heart Association Class III or IV, unstable angina pectoris, serious cardiac arrhythmias.
  * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 3 months before the first dose.
  * QTc prolongation defined as a QTcF > 500 ms.
  * Known congenital long QT.
  * Left ventricular ejection fraction < 55%.
  * Uncontrolled hypertension defined as ≥ 140/90 as assessed from the mean of three consecutive blood pressure measurements taken over 10 minutes.
* Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the drug through a feeding tube], social/psychological issues, etc.)
* HIV infection with a detectable viral load within 6 months of the anticipated start of treatment.

  --Note: Subjects on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and TB testing in line with local practice), hepatitis B (positive HBV surface antigen (HBsAg) result), or hepatitis C.

  --Note: Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to investigational product (IP) or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.7.2. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Rate of pathologic response rate (pCR, mCR/nCR, or pPR) at the time of surgery. | 2 months
  Assess the pathologic response rate (pRR) at the time of surgery after two doses of neoadjuvant Ipilimumab and Nivolumab for patients that have recurred while receiving/recently completed adjuvant anti-PD1 therapy.

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE, version 5.0), seriousness, duration, and relationship to study treatment. | 2 months
  Assess the safety and tolerability of Ipilimumab and Nivolumab in the study population.
Rate of adverse events that occur within 30 days post-surgery. | 30 days
  Assess the impact of neoadjuvant ipi/nivo on morbidity of definitive surgery.
Rate of Event Free Survival (EFS). | 11 years
  Assess EFS in the study population.
Rate of Overall Survival (OS). | 11 years
  Assess OS in this study population.
Objective response rate (ORR) defined as the proportion of subjects achieving a confirmed PR and CR as defined by RECIST 1.1 prior to surgical resection. | 11 years
  Determine RECIST 1.1 response rate (confirmed CR and PR) before surgical resection and to evaluate associations between radiographic and pathologic response rate and event free survival/overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Siwen Hu-Lieskovan, PhD, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No